CLINICAL TRIAL: NCT06984770
Title: Caring for the Caregiver: A Pilot Randomized Controlled Trial (The Family Cares Trial)
Brief Title: The Family Cares Trial
Acronym: Family Cares
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Michael Goldfarb, Attending Staff, Division of Cardiology, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MP-05-2026-4603
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Family Engagement; Critical Care, Intensive Care; Patient and Family Engagement; Health Care Delivery; Family-centered Care; Pilot Study; Caregiver; Caregiver Burden; Family Caregivers
Keywords: Patient- and Family-Centered Care; Family Engagement; Critical Care; Intensive Care Unit; Person-Centered Care; Delivery of Health Care; Post-ICU; Caregivers; Family Caregiver
MeSH Terms: conditions — Caregiver Burden | interventions — Health Resources

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: Resources only (Active Comparator): Participants will be given a list of resources for emotional or psychological distress.
  Interventions: Other: Resources
- Intervention Group (Experimental): Participants assigned to the intervention group will be permitted to choose which strategy they wish to participate in. This innovative person-centered approach will ensure that family caregivers get the type of support that they want and are not arbitrarily assigned to a strategy that they are not motivated to pursue, resulting in a pragmatic, real-world approach to choice of strategy. Participants will have the choice of two strategies: 'Virtual peer support group' or 'Caregiver Support'.
  Interventions: Behavioral: Virtual peer support group intervention; Behavioral: Caregiver Support intervention; Other: Resources

INTERVENTIONS:
Behavioral: Virtual peer support group intervention — The virtual peer support group aims to improve emotional well-being, reduce isolation, and help caregivers cope by offering a safe space to share experiences and receive support from others facing similar caregiving demands.
  Arms: Intervention Group
Behavioral: Caregiver Support intervention — The caregiver support intervention is a personalized program designed to improve quality of life, reduce fatigue and caregiver burden, and build resilience.
  Arms: Intervention Group
Other: Resources — Participants will be given a list of resources to contact in case of emotional or psychological distress.

SUMMARY:
The goal of this pilot study is to learn if virtual peer support groups and strengths-based skills training can help family caregivers of ICU survivors providing ongoing support to ICU survivors after hospital discharge. The main question it aims to answer is:

- Are virtual peer support groups and/or strengths-based skills support feasible and acceptable for family caregivers of ICU survivors? Researchers will compare the intervention group (virtual peer support groups or strengths-based skills training) to the control group (no intervention) to see if the interventions improve caregiver outcomes and assess feasibility and acceptability.

Participants will:

* Participate in either virtual peer support groups or strengths-based skills training sessions (if assigned to the intervention arm).
* Provide feedback on the feasibility and acceptability of the interventions (if assigned to the intervention arm).
* Complete surveys and follow-up questionnaires (either online or by phone) to measure outcomes.

ELIGIBILITY:
Inclusion Criteria:

* (1) Family member of a person admitted to an ICU for >48 hours and survived to hospital discharge. "Family" is anyone with a biological, legal, or emotional relationship with the patient and whom the patient wants involved in their care
* (2) Planned or current part or full-time caregiver of the ICU survivor
* (3) Age ≥ 18 years
* (4) Within 6 months of ICU survivor's hospital discharge.

Exclusion Criteria:

* (1) Another family member participating in the study
* (2) Inability to communicate in English or French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Caregiver Burden - The Zarit Burden Interview-12 (ZBI-12) - 3 months | 3 months post-enrollment or post intervention initiation
  A 12-item self-report tool that has been validated for measuring the level of caregiver burden related to care provision. Each item in the ZBI-12 is scored on a five-point Likert scale from 0 to 4 (0=never to 4=nearly always). Summed scores range from 0-48, with greater scores representing greater feelings of burden.

SECONDARY OUTCOMES:
Caregiver Burden - The Zarit Burden Interview-12 (ZBI-12) - 6 months | 6 months post-enrollment or post intervention initiation
  A 12-item self-report tool that has been validated for measuring the level of caregiver burden related to care provision. Each item in the ZBI-12 is scored on a five-point Likert scale from 0 to 4 (0=never to 4=nearly always). Summed scores range from 0-48, with greater scores representing greater feelings of burden.
Multidimensional Scale of Perceived Social Support (MSPSS) - 3 months | 3 months post-enrollment or post intervention initiation
  A 12-item self-report tool that has been validated for measuring perceived social support from family, friends and significant others. Each item is scored on a likert scale from 1-7, where 1= Very strongly disagree, and 7= very strongly agree. Total scores range from 12 to 84, where a score of 12-35 could be considered low support; a score of 33 to 60 could be considered moderate support; a score from 61 to 84 could be considered high support.
Multidimensional Scale of Perceived Social Support (MSPSS) - 6 months | 6 months post-enrollment or post intervention initiation
  A 12-item self-report tool that has been validated for measuring perceived social support from family, friends and significant others. Each item is scored on a likert scale from 1-7, where 1= Very strongly disagree, and 7= very strongly agree. Total scores range from 12 to 84, where a score of 12-35 could be considered low support; a score of 33 to 60 could be considered moderate support; a score from 61 to 84 could be considered high support.
Patient Health Questionnaire-9 (PHQ-9) - 3 months | 3 months post-enrollment or post intervention initiation
  A 9-item self-reported tool to quantify depression symptoms and monitor severity. Each item is scored using a 4-point Likert scale ranging from 0-3 (not at all=0, several days=1, more than half the days=2, and nearly every day=3). The total score can range from 0 to 27, where a total score of 0-4 indicates minimal to no depression, 5-9 indicates mild depression, 10-14 indicates moderate depression, 15-19 indicates moderately severe depression, and 20-27 indicates severe depression.
Patient Health Questionnaire-9 (PHQ-9) - 6 months | 6 months post-enrollment or post intervention initiation
  A 9-item self-reported tool to quantify depression symptoms and monitor severity. Each item is scored using a 4-point Likert scale ranging from 0-3 (not at all=0, several days=1, more than half the days=2, and nearly every day=3). The total score can range from 0 to 27, where a total score of 0-4 indicates minimal to no depression, 5-9 indicates mild depression, 10-14 indicates moderate depression, 15-19 indicates moderately severe depression, and 20-27 indicates severe depression.
Post-traumatic stress (IES-Revised) - 3 months | 3 months post-enrollment or post intervention initiation
  The IES-Revised is a 22-item questionnaire that has been validated and is widely used for measuring post-traumatic stress symptoms and yields a total score ranging from 0 to 88 and subscale scores for the Intrusion, Avoidance, and Hyperarousal subscales. Items are rated on a 5-point scale ranging from 0 (not at all) to 4 (extremely). High scores indicate greater severity of PTSD.
Post-traumatic stress (IES-Revised) - 6 months | 6 months post-enrollment or post intervention initiation
  The IES-Revised is a 22-item questionnaire that has been validated and is widely used for measuring post-traumatic stress symptoms and yields a total score ranging from 0 to 88 and subscale scores for the Intrusion, Avoidance, and Hyperarousal subscales. Items are rated on a 5-point scale ranging from 0 (not at all) to 4 (extremely). High scores indicate greater severity of PTSD.
Insomnia Severity Index (ISI) - 3 months | 3 months post-enrollment or post intervention initiation
  A 7-item self-report questionnaire that has been validated for measuring the nature, severity, and impact of insomnia. Responses on each item can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia. Total score ranges from 0-28, and can be interpreted as follows: a total score of 0-7 indicates "no clinically significant insomnia," 8-14 indicates "subthreshold insomnia," 15-21 indicates "clinical insomnia (moderate severity)," and 22-28 indicates "clinical insomnia (severe).
Insomnia Severity Index (ISI) - 6 months | 6 months post-enrollment or post intervention initiation
  A 7-item self-report questionnaire that has been validated for measuring the nature, severity, and impact of insomnia. Responses on each item can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia. Total score ranges from 0-28, and can be interpreted as follows: a total score of 0-7 indicates "no clinically significant insomnia," 8-14 indicates "subthreshold insomnia," 15-21 indicates "clinical insomnia (moderate severity)," and 22-28 indicates "clinical insomnia (severe).
Quality of life (EuroQOL-5D-5L score) - 3 months | 3 months post-enrollment or post intervention initiation
  The EuroQOL-5D-5L is a 5-item questionnaire that has been validated and is widely used for measuring health-related quality of life. Each dimension has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). The scores are combined to generate a single index value for overall health status. EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state
Quality of life (EuroQOL-5D-5L score) - 6 months | 6 months post-enrollment or post intervention initiation
  The EuroQOL-5D-5L is a 5-item questionnaire that has been validated and is widely used for measuring health-related quality of life. Each dimension has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). The scores are combined to generate a single index value for overall health status. EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state
Connor-Davidson Resilience Scale-10 (CD-RISC 10) - 3 months | 3 months post-enrollment or post intervention initiation
  A 10-item self-report tool that has been validated for measuring resilience. Each item is scored on a 5-point Likert scale (0 = "not true at all" to 4 = "true nearly all the time"). The total score ranges from 0 to 40, with higher scores indicating greater resilience.
Connor-Davidson Resilience Scale-10 (CD-RISC 10) - 6 months | 6 months post-enrollment or post intervention initiation
  A 10-item self-report tool that has been validated for measuring resilience. Each item is scored on a 5-point Likert scale (0 = "not true at all" to 4 = "true nearly all the time"). The total score ranges from 0 to 40, with higher scores indicating greater resilience.

OTHER OUTCOMES:
FAM-Activate (FAM-A) | completed at enrolment in the study
  The FAM-Activate (FAM-A) tool is a self-administered 4-item questionnaire that assesses an individual's current activation. FAM-A uses a five-point Likert scale ranging from 1 (strongly agree) to 5 (strongly disagree), and scale results are changed to a 0-100 scoring system, with higher scores indicating greater activation. Activation refers to the knowledge, skills, and confidence of a family member.
FAMily Engagement (FAME) | completed at enrolment in the study
  The FAMily Engagement (FAME) tool is a self-administered 12-item questionnaire that assesses an individual's current engagement practice. FAME uses a five-point Likert scale ranging from 1 (strongly agree) to 5 (strongly disagree), and scale results are changed to a 0-100 scoring system, with higher scores indicating greater engagement in care. The following subdomains are evaluated: engagement perception, family presence, communication, education, decision-making, care contribution, and family needs. FAME includes the following engagement domains: family presence, family needs, communication and education, decision making, and direct care. FAME also captures the following family-centered care principles: dignity and respect, information sharing, participation, and collaboration.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Goldfarb, MD, MSc, Principal Investigator — Lady Davis Institute, McGill University, Jewish General Hospital
Locations (2):
- Canada (2):
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No